CLINICAL TRIAL: NCT02199171
Title: A Phase I Dose-escalation and Pharmacokinetic Study of Hyperthermic Intraoperative Intraperitoneal Chemotherapy (HIPEC) Carboplatin at the Time of Cytoreductive Surgery for the Initial Treatment in Patients With Advanced Ovarian, Fallopian Tube, and Peritoneal Carcinomas.
Brief Title: Heated Carboplatin in Treating Patients With Stage II-IV Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Krishnansu, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 13-54 HS# 2014-1188; 2014-1188 (Other: University of California, Irvine)
Record Dates: First submitted 2014-07-16; First posted 2014-07-24 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: FIGO Stage IIC-IV Ovarian Carcinoma; Fallopian Tube Carcinoma; Peritoneal Carcinoma
Keywords: hyperthermic intraoperative intraperitoneal chemotherapy (HIPEC) carboplatin; intraperitoneal (IP) chemotherapy; cytoreductive surgery
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Carboplatin; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIPEC carboplatin (Experimental): Patients receive hyperthermic carboplatin intraperitoneally over 60 minutes during the planned surgical cytoreductive procedure.
  Doses as appropriate for assigned dose level in 500 cubic centimeters (cc)
  Interventions: Drug: carboplatin

INTERVENTIONS:
Drug: carboplatin — Given via HIPEC
  Other Names: (SP-4-2)-diammine[1,1-cyclobutanedicarboxylato(2--)-O,O']platinum, 1,1-cyclobutanedicarboxylic acid platinum complex; 19314; 241240; 41575-94-4; Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; cis-diammine(1,1-cyclobutanedicarboxylato) platinum(II); cis-diammine(cyclobutane-1,1-dicarboxylato)platinum; cis-diammine(cyclobutanedicarboxylato)platinum II; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; platinum; diammine(1,1-cyclobutanedicarboxylato(2-))-; (SP-4-2); Platinwas; Ribocarbo

SUMMARY:
This phase I trial studies the side effects and best dose of heated carboplatin given into the abdomen at the time of surgery in treating patients with stage II-IV ovarian, fallopian tube, or peritoneal cancer. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Heating oxaliplatin and infusing it directly into the area around the tumor during surgery may kill more tumor cells.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the maximum tolerated dose (MTD) of carboplatin given as HIPEC for primary treatment of women with advanced ovarian, peritoneal, and fallopian tube cancers.

Secondary Objectives:

1. To determine the dose limiting toxicities of HIPEC carboplatin.
2. To describe the pharmacokinetic profile of HIPEC carboplatin.
3. To quantify changes in tissue temperature during HIPEC and compare to conventional temperature measures (esophageal and bladder).
4. To describe the extent of thermal damage and DNA platinum adduct formation in tissues resulting from HIPEC carboplatin.

OUTLINE: This is a dose escalation study.

Patients receive hyperthermic carboplatin intraperitoneally over 60 minutes during the planned surgical cytoreductive procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed, known or highly suspected advanced (International Federation of Gynecology and Obstetrics [FIGO] stage II-IV) ovarian, primary peritoneal, or fallopian tube cancer, scheduled for primary or interval cytoreductive surgery
* If the patient has received pre-operative neoadjuvant chemotherapy, evidence of response must be documented by at least one of the following: decline in serum carcinoma antigen (CA)125 level, at least a 30% decrease in the sum of the longest diameter of target lesions on radiographic imaging, or resolution of ascites or pleural effusion(s)
* Women of all races and ethnic groups are eligible for this trial
* Gynecologic Oncology Group (GOG) performance status =< 2
* Leukocytes >= 3,000/microliter (mcL)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT))/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Albumin >= 2.5 mg/dL
* Patients for whom the diagnosis of high-grade serous or undifferentiated carcinoma of ovarian, peritoneal, or fallopian tubal origin is confirmed at surgery
* Surgery achieves either no gross residual disease or optimal cytoreductive status defined as no single lesion measuring more than 1 cm in its greatest diameter (this protocol calls for the intentional delay in resection of up to 3 tumors per patient until the HIPEC procedure is complete; the surgeon will identify these tumors as easily resectable from a technical and safety aspect)
* Patients must be stable from cardiopulmonary and hemodynamic standpoints to continue with prolonged surgery and anesthesia
* Provision of written informed consent

Exclusion Criteria:

* Patients receiving neo-adjuvant chemotherapy whose disease has progressed following at least 3 cycles, defined by at least one of the following: clinical deterioration (new or worsening of existing ascites, carcinomatous ileus, malignant bowel obstruction, declining performance status), new lesion(s) or increase in maximal diameter of > 20% of the two largest target lesions, rising CA-125 (an increase of at least 10% of baseline value that increases over 3 values obtained every 21 days)
* Cardiac or pulmonary conditions that preclude aggressive cytoreductive surgery
* Patients found to have non-gynecologic, uterine, or breast primary at surgery
* Patients with gynecologic malignancy of low-grade serous or borderline histology
* Patients with sub-optimal resection (any single tumor larger than 1 cm)
* Patients with core body temperature > 37 degrees Celsius (C) at completion of cytoreductive surgery and prior to HIPEC
* Patients who are receiving other investigational therapeutic agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of HIPEC carboplatin | Up to 30 days after study treatment
  MTD of HIPEC carboplatin, defined as the dose level with < 2 patients of 6 experiencing dose-limiting toxicities, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
  Identified using the continual reassessment method.

SECONDARY OUTCOMES:
Disease control rates, scored according to Response Evaluation Criteria in Solid Tumors criteria and consist of complete response, partial response, and stable disease | Up to 1 year
1-year overall survival (OS) rate | At 1 year
  For 1-year OS rate, death events will be recorded. One-year OS rate will be defined by the number of participants alive 1 year from the time of study entry.
Incidence of adverse events assessed using Common Toxicity Criteria version 4.0 | Up to 30 days after study treatment
  Participants who receive any amount of study drug will be evaluable for toxicity.
Change in pharmacokinetic profile of HIPEC carboplatin | Baseline and at 5, 15, 30, 45, and 60 minutes
  Median, range, and interquartile range will be calculated and reported for the amount of carboplatin absorbed from the perfusate, the rate of drug absorption from the peritoneal cavity into the systemic circulation, the 0-to-60 minute area under the curve (AUCs) for peritoneal and plasma platinum concentration curves, the total body clearance, the 0-to-24 hour AUC for filterable platinum in the plasma, and regional advantage. Estimates of population averages will be calculated and reported using 95% confidence intervals.
Changes in tissue temperature during HIPEC compared to conventional temperature measures (esophageal and bladder) | Baseline to after completion of HIPEC
  Measured at in situ tumor sites and at esophageal and bladder tissue (controls). Median, range and interquartile range will be calculated and reported for mean and peak temperature. Average within-patient paired differences of mean temperature will be summarized descriptively. Estimates of the population average difference in mean temperature between tumor and control tissue will be calculated and reported with 95% confidence intervals. Frechet or type-II extreme value distributions will be used to model the peak temperature as measured in tumor sites.
Extent of DNA platinum adduct formation in tissues resulting from HIPEC carboplatin | After HIPEC but before the subject leaves the operating room (up to 2 hours)
  Platinum levels will be measured by inductively coupled plasma mass spectrometry (ICP-MS). Median, range and interquartile range will be calculated and reported for platinum levels per tumor wet weight and per tumor volume. Estimates of population average platinum level will be calculated and reported with 95% confidence intervals as based on measured values or transformed values and the normal approximation.
Thermal damage in tissues resulting from HIPEC carboplatin | After HIPEC but before the subject leaves the operating room (up to 2 hours)
  A linear model will be calculated and reported for the regression of log-transformed total depth of destruction on per-patient mean temperature as measured during perfusion at in-situ tumor sites.

CONTACTS AND LOCATIONS:
Overall Officials: Krishnansu Tewari, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No